CLINICAL TRIAL: NCT02563444
Title: Interest in Using Ultrasound Fusion in Percutaneous Interventional Radiology
Acronym: ECHOFUSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-A00413-44
Record Dates: First submitted 2015-09-28; First posted 2015-09-30 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tissular Lesion
Keywords: Diagnostic (Biopsy) or Therapeutic Procedure (Infiltration, Ablation)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound fusion guiding system (Experimental)
  Interventions: Device: Ultrasound fusion guiding system - TUS A-500 (Aplio 500)

INTERVENTIONS:
Device: Ultrasound fusion guiding system - TUS A-500 (Aplio 500)

SUMMARY:
The investigators want to evaluate the accuracy of an ultrasound fusion guiding system in the positioning of a needle (here the accuracy is evaluated with a 22G spinal needle), by comparing the path indicated by the ultrasound fusion (virtual line) and the path actually obtained on the control CT scan (real line).

Compared with ultrasound guidance alone or CT scan alone, the results are expected to be more accurate, saving time and irradiation (not evaluated here).

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* male or female
* women of childbearing potential should use effective contraceptive measures and indicate the date of the last menstrual
* Patient requiring the use of computed tomographic guidance to perform a diagnostic (biopsy) or therapeutic procedure (infiltration, ablation) on a mobile organ
* patient signed an informed consent

Exclusion Criteria:

* Contraindications to the use of X-rays (pregnancy)
* Patients using vital electronic devices (eg: pacemaker or defibrillator)
* Subject under judicial protection
* Subject under tutorship or curatorship
* Inability to give informed informations (subject in emergency situations, comprehension difficulties of the subject, ...)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Measure of the averages (m) errors of the coordinates in the three planes of space, between the virtual and the real line of the spinal needle (comparison of ultrasound fusion data with control CT scan data achieved once the spinal needle is placed) | time of the procedure

SECONDARY OUTCOMES:
distance between the center of the target and the extension of the spinal needle (perpendicular line to this projection through the center of the lesion) | time of the procedure
overall satisfaction score | time of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Afshin GANGI, MD, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- Nouvel Hôpital Civil, Strasbourg, Alsace, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bing F, Vappou J, Breton E, Enescu I, Garnon J, Gangi A. Accuracy of a CT-Ultrasound Fusion Imaging Guidance System Used for Hepatic Percutaneous Procedures. J Vasc Interv Radiol. 2019 Jul;30(7):1013-1020. doi: 10.1016/j.jvir.2018.11.034. Epub 2019 Mar 25. PMID 30922795
- [Result] Garnon J, Koch G, Tsoumakidou G, Caudrelier J, Chari B, Cazzato RL, Gangi A. Ultrasound-Guided Biopsies of Bone Lesions Without Cortical Disruption Using Fusion Imaging and Needle Tracking: Proof of Concept. Cardiovasc Intervent Radiol. 2017 Aug;40(8):1267-1273. doi: 10.1007/s00270-017-1638-9. Epub 2017 Mar 29. PMID 28357575